CLINICAL TRIAL: NCT01556256
Title: Music Video for AYA-Parent Communication and Resilience
Brief Title: Music Therapy Video Development in Improving Communication, Emotional Distress, and Recovery in Adolescents/Young Adults Undergoing Treatment for High-Risk Cancer and Their Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ANUR1131; NCI-2012-00682 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000726664; COG-ANUR1131; ANUR1131 (Other: Children's Oncology Group); COG-ANUR1131 (Other: DCP); ANUR1131 (Other: CTEP); R01CA162181 (NIH); U10CA095861 (NIH); UG1CA189955 (NIH)
Record Dates: First submitted 2012-03-15; First posted 2012-03-16 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (TMV) (Experimental): See detailed description.
  Interventions: Procedure: Music Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (TMV+P) (Experimental): See detailed description.
  Interventions: Other: Caregiver-Related Intervention or Procedure; Procedure: Music Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Caregiver-Related Intervention or Procedure — Undergo TMV+P
  Arms: Arm II (TMV+P)
Procedure: Music Therapy — Undergo TMV
  Arms: Arm I (TMV)
Procedure: Music Therapy — Undergo TMV+P
  Arms: Arm II (TMV+P)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized trial studies how well music therapy and parents' education work in improving communication, emotional distress, and recovery in adolescents/young adult patients undergoing treatment for high-risk cancer and their parents. Making a music therapy video may improve communication, emotional distress, and recovery in younger patients undergoing treatment for cancer. It is not yet known whether music therapy and counseling for parents is more effective than information handouts for parents in improving communication and emotional distress in patients undergoing treatment for cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the efficacy of a Therapeutic Music Video (TMV) intervention with a Therapeutic Music Video plus Parent (TMV+P) intervention on outcomes for adolescents/young adults (AYA) undergoing treatment for high-risk cancer.

II. Compare the efficacy of a TMV intervention with a TMV+P intervention on outcomes for parents of AYA with high-risk cancer.

III. Determine relationships of parent distress and parent perceived family environment with AYA outcomes using a mixed methods approach. (exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to age in years (11-13 vs 14-17 vs 18-24). Parents are randomized to 1 of 2 intervention arms.

ARM I (TMV, low-dose parent): AYA patients undergo 60-minute sessions, delivered in a private setting during outpatient clinic visits or hospitalizations, within a 6-8 weeks period with board-certified music therapists. The music therapists help patients in brainstorming and lyric writing, singing and creatively exploring how AYA lyrics and structure of the selected music fit together, recording their song with a digital accompaniment track, completing video layout worksheets (determining the contents of the video), taking and gathering photos or making drawings for the video, and viewing clip art and pictures on a computer. The music therapist then digitally formats, compiles, and transfers the AYA-developed music video to a DVD. When completed, the therapist shares the video with the AYA and offers the option of having a video "premiere." AYAs who choose a premiere select a date and time for the viewing and identify individuals they wish to attend (family, friends, healthcare professionals). After the viewing, AYAs receive a copy of their DVD to keep. Parents' presence and involvement during all sessions are directed by the AYAs. Parents receive 2 sessions over 15-60 minutes with a trained study team. During the first session, parents receive handouts of helpful website resources that have specific information to help parents support their AYAs. Team members also assure that parents know how to assess the sites. During the second session, parents receive audio-recorded, telephone-based contact by a trained nurse who asks them questions focusing on the content available on the provided website. The trained nurse also answers any questions parents may have.

ARM II (AYA TMV +P): AYA patients receive intervention as patients in arm I. Parents receive 3 tailored 60-minute sessions with a trained nurse intervener. Sessions are recorded to make sure study nurse delivers the sessions according to the study protocol. Study nurse provides support information to parents using the Robb's Contextual Support Model, including Managing the Chaos: Self Care as the First Step to Caring for Your AYA, Relationship Support: How to Listen to and Encourage Your AYA to Talk; and Strategies for AYA Autonomy Support: Understanding AYA's Ways of Coping. Session 3 content is also based on the Resilience in Illness model. Sessions are also tailored to parents' needs, skills practice and/or role playing, and reflection on and reinforcement of learning. Parents receive written materials on tips and prescribed skills practice plans. AYA and parents complete questionnaires including Illness-Related Distress, Defensive Coping, Spiritual Perspective, Social Integration, Family Environment questionnaires, Hope-Derived Meaning, Self-Transcendence, Positive Coping, Resilience, Parent Distress, and Quality of Life at baseline, at 2 weeks after final session, and then at 90 days after final intervention session. Medical background, intensity of treatment rating scale, and family demographics are also collected.

ELIGIBILITY:
Inclusion Criteria:

* AYA has initial or relapsed cancer diagnosis and is actively on treatment and will continue to be on treatment long enough to complete the intervention and evaluation (4 to 6 weeks)
* AYA meets at least 1 of 3 criteria indicating potentially high palliative care or end-of-life needs:

  * Any high-risk cancer (i.e., metastatic or stage IV)
  * Receiving moderate- to high-intensity chemotherapy during 3-5 consecutive days in an in- or out-patient setting
  * A diagnosis with an estimated 5-year event-free survival of < 50%
* AYA is able to participate in sessions as evaluated by the Karnofsky/Lansky score of 50% or greater
* One consistent parent is willing and available to participate in all parent and evaluation sessions
* AYA is not married and has no children
* AYA and parent are able to read, understand, and speak English

Exclusion Criteria:

* Cancers not usually occurring in childhood/adolescent or young adult populations, such as lung or prostate cancer
* Cognitive impairments that would make it difficult for AYA/parents to participate in the intervention or complete questionnaires (determination in consultation with attending physician, oncologist, and, for adolescents below age 18, the parents)

Ages: 11 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2012-04-23 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
AYA illness-related distress measured by the Mishel Uncertainty in Illness Scale and the McCorkle Symptom Distress scale | Up to 90 days
  The MPLUS software will be used to perform latent variable analysis of covariance (ANCOVA) to account for measurement error and to reduce the number of comparisons.
AYA defensive coping measured by the Jalowiec Coping Scale-Revised | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
AYA spiritual perspective measured by the Reed Spiritual Perspective Scale | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
AYA social integration measured by the Perceived Social Support-Family scale, the Perceived Social Support-Friends scale, and the Perceived Social Support-Health Care Providers | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
AYA family environment measured by the Family Adaptability and Cohesion Scale II | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
AYA family environment measured by the Parent-Adolescent Communication scale | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
AYA family environment measured by the Family Strengths Scale | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
AYA positive coping measured by the Jalowiec Coping Scale-Revised | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
AYA hope-derived meaning measured by the Herth Hope Index | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
AYA self-transcendence measured by the Reed Self-Transcendence scale | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
AYA resilience measured by the Nowotny Confidence subscale, the Haase Resilience in Illness Scale, and the Index of Well-Being | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
Parental distress measured by the Perceived Stress Scale, the Profile of Mood States-Short Form, and the Spielberger's State-Trait Anxiety Inventory-State Component | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
Parent family environment measured by the Family Adaptability and Cohesion Scale | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
Parent family environment measured by the Parent-Adolescent Communication scale | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
Parent family environment measured by the Family Strengths Scale | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
Parent family environment measured by the Perceived Social Support-Health Care Providers | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.
Parent quality of life measured by the Index of Well-being | Up to 90 days
  The MPLUS software will be used to perform latent variable ANCOVA to account for measurement error and to reduce the number of comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Joan E Haase, Principal Investigator — Children's Oncology Group
Locations (8):
- United States (8):
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Children's Healthcare of Atlanta - Scottish Rite, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas